CLINICAL TRIAL: NCT05328414
Title: Steroid Loaded Intranasal Films as a Local Treatment of Anosmia
Brief Title: Preparation and Characterization Intranasal Film Loaded With Steroid as a Local Treatment of Anosmia in Compare to Insulin Intranasal Film
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Principal Investigator, Soad Ali, Clinical professor, Deraya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pinsfilm
Record Dates: First submitted 2022-03-27; First posted 2022-04-14 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Smell Loss
MeSH Terms: conditions — Anosmia | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Drug: Prednisolone
- steroid based intranasal film (Experimental)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — intranasal fast dissolving film to be applied intranasal. it contains 0.005 mg Presdnisolone

SUMMARY:
This study is a growing step of phase I study published on March 2021. The study was implicated on Minia university on small scale of patient (20) to investigate the impact of insulin as fast dissolving films for intranasal delivery to treat anosmia in post COVID-19 infections. this record will modify the first formulation by addition certain concentration of steroid.

ELIGIBILITY:
Inclusion Criteria:

* All patients' adults aged from 18 years to 50 will included in the study.
* A confirmed case (positive PCR), recovered/discharged (2 negative PCR),
* suffering from sudden recent anosmia or hyposmia with or without loss of taste.

Exclusion Criteria:

1. Patients with chronic sinusitis.
2. Patients with acute allergic rhinitis.
3. Patients' nasal polyposis
4. Patients with history of nasal surgery, severe head trauma or any medical condition that may affect sense of smell.
5. Patient poly morbidities or poly pharmacy.
6. Elder, pregnant, or nursing woman.
7. Patients with chronic diseases.
8. Autoimmune diseases.
9. Patient suffering end organ problems.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Smell restoring | three week
  Discrmination test; to recogonize the odd odor three times trial
Smell restoring | three week
  Sniffs test; to recogonize the first concentration he could identify

SECONDARY OUTCOMES:
inflammation | three weeks
  to measure the extent of inflammation the reddness and size

CONTACTS AND LOCATIONS:
Locations (1):
- Soad A. Mohamad, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No